CLINICAL TRIAL: NCT05683275
Title: Short and Long Term Effects of Instrument Assisted Soft Tissue Mobilization and Extracorporeal Shock Wave Therapy in Individuals With Lateral Epicondylitis
Brief Title: Short and Long Term Effects of IASTM and ESWT Therapy in Individuals With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KaratayUH6
Record Dates: First submitted 2022-12-28; First posted 2023-01-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-12

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral epicondylitis; pain; function; grip strength
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IASTM (Experimental): In addition to the home exercise program application, IASTM application will be made for 4 weeks. IASTM will be applied to the affected extremity twice a week for 4 weeks, in total 8 sessions. Participants will be asked to sit comfortably in a chair with back support. IASTM will be applied to the wrist extensor muscles of the participants for 90 seconds in the position where the muscle is tense, with a frequency of 60 beats per minute (Cheatham et al., 2019). The instruments will be applied to the soft tissue at 30º-60º angles, using vaseline as an intermediate, with a multidirectional "stroking" movement.
  Interventions: Other: IASTM
- ESWT (Experimental): ESWT will be applied to the affected elbow two days a week for 4 weeks, a total of 8 sessions, each session 2000 shock 10 Hz frequency, 2.5 bar intensity point and circumferential application. Ultrasound gel will be used as an intermediate in the application. No anesthetic substance will be used before and after the application. Cold applications will be recommended for those who have pain after the application.
  Interventions: Other: ESWT
- Home Exercise (Experimental): Static stretching and eccentric strengthening exercises specific to the forearm muscles will be taught and they will be asked to perform 2 sets (morning-lunch-evening) 10 repetitions per day, 5 days a week, for 4 weeks. For strengthening exercises, all patients will be asked to use green (medium resistance) elastic bands, hold them in a tense position for 10 seconds, let them back passively, and rest for 1 minute between sets. In the stretching exercise, they will be asked to stay in the most tense position for 30-45 seconds and rest for 30 seconds between stretching. In case of a painful situation, they will be asked to be informed about their information.
  Interventions: Other: Home Exercise

INTERVENTIONS:
Other: IASTM — IASTM will be applied to the affected extremity twice a week for 4 weeks, in total 8 sessions. Participants will be asked to sit comfortably in a chair with back support. IASTM will be applied to the wrist extensor muscles of the participants for 90 seconds in the position where the muscle is tense, with a frequency of 60 beats per minute.
  Arms: IASTM
Other: ESWT — ESWT will be applied to the affected elbow two days a week for 4 weeks, a total of 8 sessions, each session 2000 shock 10 Hz frequency, 2.5 bar intensity point and circumferential application.
  Arms: ESWT
Other: Home Exercise — Special static stretching and eccentric strengthening exercises for the forearm muscles will be taught and they will be asked to perform 2 sets (morning-lunch-evening) 10 repetitions per day, 5 days a week, for 4 weeks.
  Arms: Home Exercise

SUMMARY:
Pain, decreased grip strength, and loss of function are observed in individuals with lateral epicondylitis. The aim of this study is to investigate the effects of ESWT and IASTM applications on pain, grip strength and function in individuals with lateral epicondylitis.

DETAILED DESCRIPTION:
The study will be carried out on volunteers after the approval of the ethics committee. Before the research, individuals and / or their relatives will be informed about the purpose and content of the study. Participants will be randomly divided into three groups: IASTM, ESWT and home exercise group. In addition to home exercise, IASTM and ESWT groups will be given 2 sessions per week for 4 weeks. Pain, grip strength and functionality of the participants will be evaluated before the application, after 4 weeks of application and 4 weeks after the end of the application.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with chronic LET by a physician
* visual analog scale (VAS) pain score ≥ 3

Exclusion Criteria:

* any accompanying pathology in the wrist and forearm, such as a fracture or dislocation of the elbow;
* treatment with corticosteroid injections in the past 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain assessed by Visual Analog Scale. | Baseline, 4 weeks
  Pain will be evaluated with Visual Analog Scale. 0 means no pain, 10 means unbearable pain.

SECONDARY OUTCOMES:
Grip strength | Baseline, 4 weeks
  Grip strength will be evaluated with Hand Dynamometer
Function assessed by Patient-rated Forearm Evaluation Questionnaire | Baseline, 4 weeks
  Function will be evaluated with Patient-rated Forearm Evaluation Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)